CLINICAL TRIAL: NCT03711513
Title: Core Elements of Cognitive Behavioural Therapy in Treating Speech Anxiety in Youth: Facing Fears by Focussing on Behaviour, Body, or Mind?
Brief Title: Facing Fears by Focussing on Behaviour, Body, or Mind?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Rachel de Jong, MSc, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL60377.042.16
Record Dates: First submitted 2018-07-30; First posted 2018-10-18 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Social Anxiety
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure only (Experimental): Psycho-education (PE) (plus homework) + 4 x Exposure (EX) (plus homework): 20 participants will receive four exposure group sessions after the psycho-education session. In the four sessions they will move up in their fear hierarchy by practicing public speaking/performance tasks.
  Interventions: Behavioral: Cognitive behavioral therapy
- Cognitive restructuring plus exposure (Experimental): PE (plus homework) + Cognitive Restructuring (CR) (plus homework) + CR (plus homework) + EX (plus homework) + EX: 20 participants will receive two cognitive restructuring group sessions after the psycho-education session. In these two session they will practice identifying dysfunctional cognitions and formulating more functional (alternative/helping) cognitions. After the cognitive sessions they will receive two exposure group sessions. In these two sessions they will move up in their fear hierarchy by practicing public speaking/performance tasks.
  Interventions: Behavioral: Cognitive behavioral therapy
- Relaxation plus exposure (Experimental): PE (plus homework) + Relaxation (RE) (plus homework) + RE (plus homework) + EX (plus homework) + EX: 20 participants will receive two relaxation exercises group sessions after the psycho-education session. In these two session they will practice muscle relaxation and breathing exercises. After the relaxation sessions they will receive two exposure group sessions. In these two sessions they will move up in their fear hierarchy by practicing public speaking/performance tasks.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — All conditions start with a psycho-education session (PE). Subsequently, participants in condition A follow four exposure sessions (EX). Participants in condition B follow two cognitive restructuring (CR) followed by two exposure sessions. Participants in condition C follow two relaxation exercises sessions (RE) followed by two exposure sessions. All sessions will take place at their school in a group of five to eight adolescents (week 9,10,11,12,13,14). The sessions will be provided by a psychologist who receives training and supervision by a certified CBT therapist. The psychologist is assisted by a master student in psychology.

SUMMARY:
Anxiety problems are a major concern of youth mental health given that the prevalence of anxiety disorders in Dutch adolescents aged 12 to 18 is approximately 10 percent. In this group, social phobia like speech or performance anxiety are among the most common. Intervention programs based on the principles of exposure-based Cognitive Behavioral Therapy (CBT) have proven to be the most effective and most applied in therapy for social anxiety among adolescents. Thus far, research has mainly focused on effectiveness of "intervention packages" consisting of multiple CBT elements (i.e., exposure plus cognitive restructuring and relaxation exercises). The most common CBT element in current intervention packages for anxiety in youth is exposure, which is often only applied after providing the child with cognitive restructuring (CR) and relaxation exercises (RE) as preparation for exposure. However, although most empirical evidence supports the value of the use of exposure, there is hardly empirical evidence for the additional value of CR or RE. In addition, it is unclear whether the combination of these elements with exposure is counterproductive compared to the use of exposure only. After all, without lengthening the treatment, the addition of CR and/or RE will leave the therapist and child with less time to spend on exposure exercises.This study proposes to evaluate the effectiveness of these three different types of CBT-elements in the treatment of speech/performance anxiety among adolescents.

DETAILED DESCRIPTION:
Objective: The primary goal of this study is to evaluate which elements add to the effectiveness of current CBT programs. Second, it will be investigated whether the effect of exposure is reduced by the addition of cognitive restructuring and relaxation exercises. In addition, it will be explored how a given element is effective (i.e., mediation), by investigating which dimension of anxiety (approach/avoidance behavior, cognitions or bodily tension) is changed by which specific element, in a group of adolescents with the performance/public speaking subtype of social phobia.

Study design: Randomized Controlled Trial with three parallel groups (intervention versus intervention versus intervention).

Study population: Adolescents aged 12 to 15 years with subclinical or higher levels of the fear of performance/public speaking subtype of social phobia.

Intervention: Adolescents will be randomly assigned to one of the three conditions based on their age, gender and severity of the social phobia. All adolescents will be offered a psycho-education session on anxiety, social phobia and exposure. Following this session either four exposure sessions (condition A) or two exposure session and two additional sessions are offered. The additional session are either two cognitive restructuring sessions (condition B) or two relaxation sessions (condition C). Each session will be given in groups consisting of five to eight participants. Every session will take up to an hour and is implemented by a psychologist assisted by a master student in psychology, who will receive training and supervision by a certified CBT therapist.

Main study parameters/endpoints (see outcome measures paragraph): The main study parameter is level of fear of performance/public speaking symptoms. Secondary study parameters are subjective level of fear, fearful cognitions, bodily tension, avoidance, coping (possible mediator variables), social phobia diagnosis, speech behavior, and self-efficacy. Tertiary study parameters are healthcare costs and quality of life (cost-effectiveness), note: cost-effectiveness is assessed for another study. Other study parameters are social phobia severity, comorbid anxiety and depression, and demographic variables (possible moderator variables); and credibility and expectancy of the treatment, treatment satisfaction, and treatment compliance (treatment characteristics).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents are aged between 12-15 years old
* Sufficient knowledge of the Dutch language
* Subclinical or higher level of the fear of performance/public speaking subtype of social phobia (SPAI-C PPF score >6 (MEAN + 1 SD); Beidel, 1996)

Exclusion Criteria:

* Absence of permission of legal guardian(s)
* Currently in treatment or receiving medication for anxiety
* Received CBT for anxiety in the past 12 months
* Past or current diagnosis of ASS/ADHD
* Different or more urgent request for help
* (Risk of) suicidality or suicidal ideation (as evidenced by checking CDI item 9 score >1 and confirmation in the ADIS interview)

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in fear of performance/public speaking symptoms | At screening (T0), 6 weeks later at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Fear of performance/public speaking symptoms will be measured by the Public Performance Factor (PPF) scale of the Social Phobia and Anxiety Inventory for Children (SPAI-C), which evaluates the somatic, cognitive and behavioural aspects of social phobia in children. This questionnaire contains 26 questions all rated on a 3-point interval scale. The PPF scale consists of 7 items. The SPAI-C has sufficient test-retest reliability and good construct, convergent and discriminative validity.

SECONDARY OUTCOMES:
Change in level of anxiety | Weekly during the five intervention weeks (T2, T3, T4, T5, T6), and one week after the last intervention sessies at post-intervention assessment (T7), and then six weeks later at follow-up assessment (T8)
  • Level of anxiety compromised of subjective level of fear, fearful cognitions, bodily tension, avoidance and coping will be measured by Visual Analogue Scales (VAS) ranging from 0-100 (ratio scale) on which the adolescent rates the following aspects of the goal situation as set in the PE session:
  * Subjective level of fear: 'I am not frightened' (0) - 'I am completely frightened' (100)
  * Fearful cognitions: 'I do not believe this at all' (0) - 'I completely believe this' (100), in which the credibility of the cognition about the feared situation as set in the PE session is rated.
  * Bodily tension: 'My body feels not tense at all' (0) - 'My body feels completely tense' (100)
  * Avoidance: 'I would never avoid this situation if I could' (0) - 'I would always avoid this situation if I could' (100)
  * Coping: 'I cannot cope with this situation at all when I encounter it' (0) - 'I can completely cope with this situation when I encounter it' (100)
Change in social phobia diagnosis | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Social phobia diagnosis in adolescents will be measured with a clinical semi-structured interview using the Anxiety Disorder Interview Schedule for Children (ADIS-IV-C). The study will only include the section of social phobia. All items offer three possible answers: yes, no or other on a nominal scale (which is chosen when the adolescent answers 'I don't know' or 'sometimes'). If the adolescent meets all three criteria for social phobia as set in the ADIS-IV, he or she will receive the social phobia diagnosis. The ADIS-IV has good test-retest reliability and concurrent validity.
Change in speech behavior | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Speech behaviour will be measured by three situational Behavioural Approach Tests (BAT) for feared and avoided situations. The test consists of a number of increasingly difficult steps in which adolescents are asked to approach a phobic situation, but are told they can stop the test at any time they wish to do so. During the BAT, individuals are asked to provide "subjective unit of disturbance scale" (SUDS 0-100 ratio scale) ratings immediately after encountering the phobic situation.
Change in self-efficacy | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Self-efficacy will be measured by the Self Efficacy Questionnaire for Children (SEQ-C). This questionnaire contains 24 questions regarding academic, social and emotional self-efficacy. Items are rated on a 5-point interval scale from 'not at all' (1) to 'very well' (5). The SEQ-C is proven to be a valid instrument with sufficient reliability.

OTHER OUTCOMES:
Change in cost-effectiveness | At pre-intervention assessment (T1) and 6 weeks after the intervention at follow-up assessment (T8)
  In addition, cost-effectiveness of the intervention will be assessed by measuring costs and quality of life (effectiveness). Measuring cost-effectiveness is not the primary goal of this research but since this study is part of a larger national project in which cost-effectiveness will also be taken into account, we consider it relevant to state here.
  * Healthcare costs will be measured by registration of costs in a cost diary based on the Trimbos Institute and Institute of Medical Technology Assessment Questionnaire on Costs Associated with Psychiatric Illness (TiC-P) and PRODISQ.
  * The EuroQol Questionaire (EQ-5D-Y youth version) will be used to establish quality of life as expressed in quality adjusted life years (QALYs).
  Healtcare costs and in quality adjusted life years (QALYs) will be combined to report cost-effectiveness.
Change in severity of the social phobia | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • The severity of the social phobia will be rated on a 0-8 interval scale by an independent psychologist on the ADIS-IV (see above). This rating is based on the level of interference, number of symptoms and general impression of the psychologist. A rating of 0, 1, 2, or 3 means no social phobia, 4 or 5 means the social phobia is mild, whereas a rating of 6, 7, or 8 means the social phobia is severe.
Change in comorbid anxiety and depression | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Given the high comorbidity of anxiety and depression in adolescents, comorbid anxiety and depression will be assessed with the Revised Child Anxiety and Depression Scale for Children (RCADS-C) consisting of 47 items. All items are rated on a 4-point interval scale from 'never' to 'always'. The RCADS has good psychometric properties.
Change in treatment credibility and expectancy | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Credibility and expectancy of the treatment are measured by the Credibility and Expectancy Questionnaire (CEQ-C). This questionnaire contains 6 items all rated on a 9-point interval scale. The psychometric properties of the scale have been qualified as good.
Change in treatment satisfaction | at pre-intervention assessment (T1), 6 weeks later at post-intervention assessment (T7), and 6 weeks later at follow-up assessment (T8)
  • Treatment satisfaction will be measured with the Service Satisfaction Scale for Children (SSS-C). Four items are rated on a 4-point interval scale ranging from 'no, definitely not' to 'yes, definitely'. The psychometric properties of the scale have been qualified as good.
Change in compliance | Weekly during the five intervention weeks (T2, T3, T4, T5, T6), and one week after the last intervention session at post-intervention assessment (T7), and then six weeks later at follow-up assessment (T8)
  • Treatment compliance will be measured using a weekly checklist in which the adolescent can state how much time they spent on the homework assignment, rated in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter de jong, Prof, Study Chair — University of Groningen; Maaike Nauta, Prof, Study Director — University of Groningen; Miriam Lommen, Dr, Study Director — University of Groningen
Locations (4):
- Netherlands (4):
  - Greijdanus College, Zwolle, Overijssel
  - RSG De Borgen Lindenborg, Leek, Provincie Groningen
  - Gomarus College, Groningen
  - CSG Augustinus, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reynolds S, Wilson C, Austin J, Hooper L. Effects of psychotherapy for anxiety in children and adolescents: a meta-analytic review. Clin Psychol Rev. 2012 Jun;32(4):251-62. doi: 10.1016/j.cpr.2012.01.005. Epub 2012 Feb 13. PMID 22459788
- [Background] Storch EA, Masia-Warner C, Dent HC, Roberti JW, Fisher PH. Psychometric evaluation of the Social Anxiety Scale for Adolescents and the Social Phobia and Anxiety Inventory for Children: construct validity and normative data. J Anxiety Disord. 2004;18(5):665-79. doi: 10.1016/j.janxdis.2003.09.002. PMID 15275945
- [Background] Silverman WK, Saavedra LM, Pina AA. Test-retest reliability of anxiety symptoms and diagnoses with the Anxiety Disorders Interview Schedule for DSM-IV: child and parent versions. J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):937-44. doi: 10.1097/00004583-200108000-00016. PMID 11501694
- [Background] Wood JJ, Piacentini JC, Bergman RL, McCracken J, Barrios V. Concurrent validity of the anxiety disorders section of the Anxiety Disorders Interview Schedule for DSM-IV: child and parent versions. J Clin Child Adolesc Psychol. 2002 Sep;31(3):335-42. doi: 10.1207/S15374424JCCP3103_05. PMID 12149971
- [Background] Koopmanschap MA. PRODISQ: a modular questionnaire on productivity and disease for economic evaluation studies. Expert Rev Pharmacoecon Outcomes Res. 2005 Feb;5(1):23-8. doi: 10.1586/14737167.5.1.23. PMID 19807557
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Brady EU, Kendall PC. Comorbidity of anxiety and depression in children and adolescents. Psychol Bull. 1992 Mar;111(2):244-55. doi: 10.1037/0033-2909.111.2.244. PMID 1557475
- [Background] Chorpita BF, Moffitt CE, Gray J. Psychometric properties of the Revised Child Anxiety and Depression Scale in a clinical sample. Behav Res Ther. 2005 Mar;43(3):309-22. doi: 10.1016/j.brat.2004.02.004. PMID 15680928
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119